CLINICAL TRIAL: NCT04175951
Title: Visual and Optical Outcomes After Bilateral Implantation of Tecnis Eyhance Versus Rayner RayOne Aspheric in Patients Undergoing Routine Cataract Surgery
Brief Title: Tecnis Eyhance Versus Rayner RayOne Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 265849
Record Dates: First submitted 2019-11-04; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Cataract Senile; Pseudophakia
Keywords: cataract; intraocular lens; intermediate vision
MeSH Terms: conditions — Pseudophakia; Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tecnis Eyhance (Active Comparator): Tecnis Eyhance hydrophobic IOL is a monofocal IOL with added advantage of slightly better unaided intermediate vision at 60 cms.
  Interventions: Device: Intraocular lens
- Rayner RayOne (Active Comparator): Rayner Rayone is a monofocal hydrophilic IOL which is not intended to give better unaided or near vision.
  Interventions: Device: Intraocular lens

INTERVENTIONS:
Device: Intraocular lens — Tecnis Eyhance is a monofocal IOL which give added intermediate vision without employing EDOF or multifocal technology and hence induces no glare and halos. Whereas monofocal IOLs such as RayOne do not give intermediate vision.

SUMMARY:
Cataract surgery involves replacing milky lens with a plastic intraocular lens. This plastic lens can be either monofocal (fixates for distance or near without glasses), extended depth of focus (EDOF)(fixates for intermediate and distance vision only without glasses) or multifocal lenses (fixates for distance, intermediate and near vision without glasses). However, EDOF and multifocal lenses are known to produce glare and halos. Tecnis Eyhance (Johnson & Johnson, USA) is a monofocal IOL which give added intermediate vision without employing EDOF or multifocal technology and hence induces no glare and halos. Whereas monofocal IOLs such as RayOne do not give intermediate vision. The objective is to assess visual and optical performance of Tecnis Eyhance versus Rayner RayOne in a prospective, randomized, comparative bilateral study. The proposed study will be the first study comparing the new technology monofocal Eyhance with conventional RayOne Rayner lens to assess the added benefits of Eyhance technology at multiple visits until 3 months after the surgery. Patients attending the clinics with cataracts will be invited to participate in this randomised study. They will be randomised to receive either Eyhance or RayOne in both eyes through surgeries performed not more than 2 weeks apart. The patients will be followed up at 1 and 3 months in the research clinic to assess the uniocular and binocular vision, spectacle prescription, a simple non-invasive scan to look at any distortions in the optics of the eye (wavefront aberrometry) and questionnaire for assessing subjective outcomes, glare and halos.

DETAILED DESCRIPTION:
Study design:

Prospective, randomised, comparative study assessing visual and optical outcomes after bilateral implantation of the new Johnson & Johnson Tecnis Eyhance versus monofocal Rayner RayOne in patients undergoing routine cataract surgery.

Methodology:

Suitable patients with cataracts in both eyes will be identified from cataract assessment clinics. They will be invited to participate in the study by the research nurse and handed over the patient information sheet and a consent form. The PI will consent the patient for the participation. If they agree to participate, they will be give the dates for their surgeries on the same day. The patients can choose to have both eyes done on the same day or two eyes within 2 weeks based on the patients convenience. If they chose to participate in the study, then the patient will have additional tests performed on the day of their cataract assessment clinic. This will take an additional 40 minutes.

On the day of the surgery, the patients will be randomised using a computer generated randomisation to receive either Tecnis Eyhance or the Rayner RayOne lens. They will have the same lens in both eyes. The patients will be invited for a research follow up visit at 1 (between 30-37 days after 2nd eye surgery) and 3 months (90-100 days after 2nd eye surgery) were simple research tests will performed including vision assessment and a scan.

At preoperative visit and 3 months the patients will be asked to fill in a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine cataract surgery with:

  * Patients with a symptomatic cataract,
  * Postoperative visual potential of 0.2 LogMAR or better
  * Corneal astigmatism ≤1.5D
  * Patients who are willing to participate in this study.

Exclusion Criteria:

* Patients under the age of 18 years,
* Eyes with any ocular comorbidity with cornea, uvea, retina or optic nerve, which may be detrimental to visual outcomes.
* Abnormal corneal topography or any other co-existing retinal or cornea conditions, astigmatism outside the study range,
* Unable to consent and unable to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-05-24 (Estimated); Study Completion 2020-10-24 (Estimated)

PRIMARY OUTCOMES:
Unaided distance visual acuity (UCDVA) (Uniocular and binocular) | 3 months postoperatively
  Uniocular and binocular uncorrected distance vision will be measured at the follow ups.
Unaided intermediate visual acuity (UIVA) (uniocular and binocular) | 3 months postoperatively
  Uniocular and binocular unaided intermediate vision will be measured at the follow ups

SECONDARY OUTCOMES:
Best corrected distance LogMAR visual acuity (CDVA) (uniocular and binocular) | 1 and 3 months postoperatively
  Uniocular and binocular best spectacle corrected distance vision will be measured at the follow ups
Manifest refraction (Diopters) | 1 and 3 months postoperatively
  Sphere, cylinder and axis of the manifest refraction will be recorded at follow ups
Defocus Curves (Diopters) | 1 and 3 months postoperatively
  Defocus curves will be plotted by adding + and - lenses to the manifest refraction
Distance correct intermediate LogMAR visual acuity (DCIVA) at 60 cm | 1 and 3 months postoperatively
  Uniocular and binocular best spectacle corrected intermediate vision will be recorded at follow ups
Wavefront aberrometry using iTrace Tracey aberrometer (Internal and total higher order and lower order aberrations)(microns) | 1 and 3 months postoperatively
  Aberrometry will be performed using iTrace machine (Tracy Technologies, USA) at all follow up visits
Quality of life outcomes assessment by the Catquest 9SF questionnaire | 1 and 3 months postoperatively
  Patients will be requested to fill a questionnaire at all follow up visits
Glare and halos questionnaire on 1-4 Likert scale | 1 and 3 months postoperatively
  (1= no glare and halos, 2= infrequent; 3 = frequent and 4 = continuous)

CONTACTS AND LOCATIONS:
Overall Officials: Mayank Nanavaty, FRCOphth,PhD, Principal Investigator — Brighton and Sussex University Hospitals NHS Trust
Locations (1):
- Brighton & Sussex University Hospitals NHS Trust, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nanavaty MA, Ashena Z, Gallagher S, Borkum S, Frattaroli P, Barbon E. Visual Acuity, Wavefront Aberrations, and Defocus Curves With an Enhanced Monofocal and a Monofocal Intraocular Lens: A Prospective, Randomized Study. J Refract Surg. 2022 Jan;38(1):10-20. doi: 10.3928/1081597X-20211109-02. Epub 2022 Jan 1. PMID 35020542